CLINICAL TRIAL: NCT02606162
Title: Outcomes of Severe Osteoporotic Fractures Hospitalized in France: the CROSS Cohort
Acronym: CROSS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hospices Civils de Lyon (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 13018; 2014-A01371-46 (Other: ANSM)
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Severe Fragility Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the outcomes of severe osteoporotic fractures hospitalized in France, the risk of incident severe fracture at 2 years and 5 years and the risk of mortality over 2 and 5 years.

DETAILED DESCRIPTION:
In France, the burden of osteoporotic fractures has been studied using cross sectional data from the French hospital national database. The availability of fracture liaison service in the main French cities allows the recruitment of a high number of these targeted patients. A large national multicenter, longitudinal, prospective cohort of patients hospitalized for severe osteoporotic fracture, the CROSS cohort ("Cohorte sur les Risques d'une OStéoporose Sévère"), in order to update data on prognosis (refracture, mortality), epidemiology and of severe osteoporotic fractures.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged above 60 years, living in France and hospitalized for severe fragility fractures in response to low-energy trauma (e.g., a fall from standing height).
* Vertebral fractures have to be confirmed by an X ray examination.
* To be eligible for the study the patient has to be included and interviewed within 12 weeks of the fracture event's diagnosis. Note : patients in guardianship or curatorship can be included in this protocol.
* Informed and free consent given and form signed and dated

Exclusion Criteria:

* Non severe fracture (for example wrist fracture), pathological fractures, high trauma fractures and per prosthetic fractures.
* Non registration with a social security scheme (holder or beneficiary).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women hospitalized for severe fragility fractures in response to low-energy trauma
Sampling Method: Non-Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Number of new severe fracture over 2 years | 2 years
  To assess the incidence of new severe fracture over 2 years in patients hospitalized for a severe fracture

SECONDARY OUTCOMES:
Number of new severe fracture over 5 years | 5 years
  To assess the incidence of new severe fracture over 5 years in patients hospitalized for a severe fracture

OTHER OUTCOMES:
Mortality rate | 2 years
  To study the risk of mortality over 2 years
Mortality rate | 5 years
  To study the risk of mortality over 5 years
Type of severe fracture | 3 months after inclusion and each year during 5 years
  * To study the role of refracture on mortality after adjustment for prefracture health status
  * To study the risk factors and phenotypes of patients hospitalized for severe fracture and to compare them between each type of severe fracture (hip,subtrochanteric, vertebrae, pelvis, humerus)
Number of patients who receive antiosteoporotic treatments and/or calcium and/or vitamin D and/or falls prevention | 3 months after inclusion and each year during 5 years
  To check the implementation of 2012 French guidelines, including on the basis on number of performed bone densitometry
Quality of life assessed by questionnaire Euroqol (EQ5D) and questionnaire (SF-36) | 3 months after inclusion and each year during 5 years
  To assess and compare the quality of life between each type of severe fracture

CONTACTS AND LOCATIONS:
Overall Officials: Karine BRIOT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No